CLINICAL TRIAL: NCT01621581
Title: A Phase 1 Open-Label Dose Escalation Safety Study of Convection Enhanced Delivery (CED) of Adeno-Associated Virus Encoding Glial Cell Line-Derived Neurotrophic Factor (AAV2-GDNF) in Subjects With Advanced Parkinson's Disease
Brief Title: AAV2-GDNF for Advanced Parkinson s Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120137; 12-N-0137
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-06-23

CONDITIONS: Parkinson's Disease
Keywords: Gene Therapy; Parkinson's Disease; Convection-Ehanced Delivery; Viral Vector
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): AAV2-GDNF vector will be delivered to each patient
  Interventions: Genetic: Convection enhanced delivery/AAV2-GDNF

INTERVENTIONS:
Genetic: Convection enhanced delivery/AAV2-GDNF — Adeno-Associated Virus Encoding Glial Cell Line-Derived Neurotrophic Factor (AAV2-GDNF) Administered via Bilateral Stereotactic Convection-Enhanced Delivery

SUMMARY:
Background:

- Glial cell line-derived neurotrophic factor (GDNF) is a chemical that may help protect and strengthen brain cells that produce dopamine. Dopamine is a chemical that affects brain function. People with Parkinson's disease (PD) have problems producing dopamine in the brain. Researchers want to see if gene transfer can help deliver GDNF into the area of the brain that is damaged by PD. The gene transferred in this study, called AAV2-GDNF, may help produce GDNF to protect the damaged brain cells.

Objectives:

- To test the safety and effectiveness of AAV2-GDNF gene transfer for advanced PD.

Eligibility:

- Individuals at least 18 years of age who have advanced PD that is not well controlled by medications.

Design:

* Participants will be in the study for about 5 years. There will be 18 outpatient study visits and a 3-day stay in the hospital. There may also be overnight stays for followup visits.
* Participants will be screened with a physical exam and medical history. Blood samples will be collected. Tests of PD symptoms and mood and memory will be given. Imaging studies will be used to find the right part of the brain to infuse the gene. The screening visit will take place up to 60 days before surgery.
* Participants will have a baseline visit about a month before the surgery. For 1 week before the baseline visit, participants will keep a diary on any motor problems. The visit will involve movement tests given before and after taking a regular dose of levodopa.
* Participants will have surgery to infuse AAV2-GDNF into the brain. The surgery will also include a lumbar puncture (spinal tap) to collect cerebrospinal fluid. After surgery, participants will recover in the hospital for at least 2 days.
* Participants will have another lumbar puncture 6 and 18 months after surgery. This will be an outpatient visit.
* Participants will have regular followup visits after the surgery. These visits will include neurological tests and movement studies. Visits with a neurosurgeon will take place 1, 2, and 4 weeks after surgery. Additional visits will take place every 3 months for the first 3 years, and then at longer intervals for up to 5 years.

DETAILED DESCRIPTION:
Objective:

While medications can temporarily alleviate the symptoms of Parkinson s disease (PD), they do not influence the degenerative process. Progressive loss of nigral dopaminergic (DA) neurons (the pathological hallmark of PD) results in progressive neurologic dysfunction and death. Glial cell line-derived neurotrophic factor (GDNF) was first identified based on its ability to promote the survival of embryonic DA neurons in vitro, and research has demonstrated beneficial effects of GDNF in animal models of PD. Preliminary clinical trials of GDNF infusions have yielded inconclusive results. Observed problems with tolerability and efficacy in these studies may have been related to the methods of delivery. Recent evidence indicates that gene transfer via direct delivery of viral vectors may represent a superior approach for the treatment of PD with GDNF.

Study population:

Twenty-four adult male and female subjects with advanced Parkinson s disease, who are candidates for surgical treatment for Parkinson s disease and who meet all Inclusion and Exclusion Criteria.

Design:

We propose a Phase 1 single-center, open-label, dose escalation, safety and tolerability study of adeno-associated virus, serotype 2 vector (AAV2) containing human GDNF complementary DNA. Bilateral catheters will be placed surgically through the skull and into the brain and the vector will be delivered by convection-enhanced delivery (CED) to both putamina (450 microliters per hemisphere) of 24 patients with advanced PD. An additional 76 subjects will be allowed for screening failures. Four escalating dose levels will be evaluated in the following dose cohorts (6 patients per cohort): Cohort 1 = 9 x 10(10)vg, Cohort 2 = 3 x 10(11)vg, Cohort 3 = 9 x 10(11)vg and Cohort 4 = 3 x 10(12)vg.

Outcome measures:

To assess the safety, tolerability, and potential clinical effects of CED of AAV2-GDNF in advanced PD patients, we will use defined clinical evaluations of PD (Unified Parkinson s Disease Rating Scale, Modified Schwab and England Activities of Daily Living scale, Hoehn and Yahr Staging, Lang and Fahn Dyskinesia Rating Scale, On-Off Patient Diary, Quality of Life, Modified Rankin Scale, Adverse Event Log and neurologic examinations), laboratory studies (hematologic, immunologic and chemistry), neuropsychological testing (Mattis Dementia Rating Scale, Beck Depression Inventory II and Parkinson Psychosis Questionnaire) and neuroimaging (magnetic resonance imaging and positron emission tomography).

ELIGIBILITY:
* INCLUSION CRITERIA:

Greater than 18 years of age.

Diagnosed with Idiopathic PD.

* Bradykinesia and
* At least 3 of the following clinical features: resting tremor, cogwheel rigidity, bradykinesia, postural reflex impairment.

The above clinical features must not be due to trauma, brain tumor, infection, cerebrovascular disease, other known neurological disease (e.g., hereditary form of PD, multiple system atrophy, progressive supranuclear palsy, striatonigral degeneration, Huntington s disease, Wilson s disease), or to known drugs, chemicals or toxicants.

Disease duration of > 5 years.

Hoehn and Yahr Stage III or IV off medication.

Disability present despite optimal antiparkinsonian medication therapy. Disability will be operationally defined as a Modified Schwab and England Activities of Daily Living Scale score of 80% or lower (during the off state).

Unified PD Rating Scale (UPDRS) (Fahn et al., 1987) total motor score greater than or equal to 30 in the defined off state.

Unequivocal responsiveness to levodopa, based on the single-dose levodopa test (as described in the CAPIT and CAPSIT guidelines). A 30% or greater improvement in the UPDRS total motor score will be required to establish unequivocal responsiveness to levodopa.

Able to provide proper Informed Consent.

Laboratory values at screening visit (unless other visit specified):

* Platelets >100,000/mm3 (transfusion independent)
* PT/PTT in normal range and INR less than or equal to 1.3 (on day prior to surgery, if taking anti-coagulants)
* Absolute neutrophil count (ANC) >1500/mm3
* Hemoglobin >10.0 g/dL (transfusion allowed)
* Aspartate aminotransferase or alanine aminotransferase <2.5 times ULN
* Total bilirubin <2.5 mg/dL
* Serum creatinine <1.5 mg/dL
* Serum anti-AAV2 total antibody titer <1000.

EXCLUSION CRITERIA:

Presence of prominent oculomotor palsy, cerebellar signs, vocal cord paresis,mean standing blood pressure below 75mmHg, pyramidal tract signs or amyotrophy.

Genetic PD disorders or with a strong family history of PD.

Presence of dementia (Montreal Cognitive Assessment less than or equal to 25).

Received an anti-dementia drug for treatment of cognitive impairment within 30 days of their screening for protocol eligibility.

Presence or history of psychosis, including if induced by anti-PD medications at doses required to improve motor symptoms.

Presence of untreated or suboptimally treated depression (Hamilton Depression Scale score >10) or a history of a serious mood disorder (i.e., requiring psychiatric hospitalization or a prior suicide attempt).

Presence of substance (drug, alcohol) abuse.

Contraindication to MRI and/or gadolinium.

Presence of normal striatal uptake on PET.

Coagulopathy, anticoagulant therapy, low platelet count, or inability to temporarily stop any antithrombotic medication.

Prior brain surgery, including GDNF, NTN, GAD, AADC therapy or deep brain stimulation.

Male or female with reproductive capacity who is unwilling to use barrier contraception throughout the study.

History of stroke or poorly controlled cardiovascular disease.

Uncontrolled hypertension or diabetes or any other acute or chronic medical condition that would increase the risks of a neurosurgical procedure.

History of malignancy (cerebral or systemic) other than treated cutaneous squamous cell or basal cell within the prior 5 years.

Clinically active infection, including acute or chronic scalp infection.

Received investigational agent within 12 weeks prior to screening.

Unable to comply with the procedures of the protocol, including frequent and prolonged follow-up.

Chronic immunosuppressive therapy (e.g., chronic steroids, TNF antagonists, chemotherapy)

Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of 4 different dose levels of AAV2-GDNF | Day 7, Day 14, 1 Month, 2 Month, 3 Month, 6 Month, 9 Month, 12 Month, 15 Month, 18 Month, 24 Month, 30 Month, 36 Month, 48 Month, 60 Month
  Treatment-related adverse events

SECONDARY OUTCOMES:
Obtain preliminary data regarding the potential for clinical responses of the 4 dose levels tested by assessing the magnitude and variability of any treatment effects (via clinical, laboratory and neuroimaging studies). | 12 Years

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Airaksinen MS, Saarma M. The GDNF family: signalling, biological functions and therapeutic value. Nat Rev Neurosci. 2002 May;3(5):383-94. doi: 10.1038/nrn812. PMID 11988777
- [Background] Backman CM, Shan L, Zhang YJ, Hoffer BJ, Leonard S, Troncoso JC, Vonsatel P, Tomac AC. Gene expression patterns for GDNF and its receptors in the human putamen affected by Parkinson's disease: a real-time PCR study. Mol Cell Endocrinol. 2006 Jun 27;252(1-2):160-6. doi: 10.1016/j.mce.2006.03.013. Epub 2006 Apr 27. PMID 16644101
- [Background] Bjorklund A, Kirik D, Rosenblad C, Georgievska B, Lundberg C, Mandel RJ. Towards a neuroprotective gene therapy for Parkinson's disease: use of adenovirus, AAV and lentivirus vectors for gene transfer of GDNF to the nigrostriatal system in the rat Parkinson model. Brain Res. 2000 Dec 15;886(1-2):82-98. doi: 10.1016/s0006-8993(00)02915-2. PMID 11119690
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS: 1. GENE THERAPY FOR PARKINSON'S, 2. PHASE 3 STUDY IN FOCUS - INTEC PHARMA'S ACCORDION PILL, 3. CLINICAL TRIALS RESOURCES. J Parkinsons Dis. 2019;9(2):251-264. doi: 10.3233/JPD-199001. No abstract available. PMID 31127735
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-N-0137.html